CLINICAL TRIAL: NCT00134901
Title: A Double-Blind, Placebo-Controlled Trial of the Effectiveness of Memantine in Treating Cocaine Dependence
Brief Title: Effectiveness of Memantine in Treating Cocaine-Dependent Individuals - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Frances R Levin, Director of Substance Use Disorder, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #4496-NIDA-12761-2; P50DA012761 (NIH)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine dependence; treatment; memantine
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Memantine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Memantine (Experimental): Memantine
  Interventions: Drug: Memantine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Memantine — Memantine
  Other Names: Memantine 40mg/day
  Arms: Memantine
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
Cocaine is one of the most widely abused drugs in the United States. Memantine is a type of drug called an NMDA receptor antagonist. It works by decreasing normal excitement in the brain. NMDA receptor antagonists have shown to reduce cocaine-induced dopamine release in animal models, as well as lessen conditioned cocaine cues. The purpose of this study is to determine the effectiveness of memantine in preventing relapse to cocaine use in cocaine dependent individuals. In addition, this study will determine whether memantine produces better results than a placebo in decreasing cocaine craving, psychological symptoms, functional impairment, and discontinuation of treatment in cocaine dependent individuals.

DETAILED DESCRIPTION:
Memantine is a non-competitive NMDA receptor antagonist that works by decreasing normal excitement in the brain. Dopamine plays a role in the rewarding and addictive properties of cocaine, however, past clinical studies have not been successful in using dopamine agonists in treating cocaine dependent individuals. Non-competitive NMDA receptor antagonists have shown to reduce cocaine-induced dopamine release in animal models and lessen conditioned cocaine cues. This study will evaluate memantine in treating cocaine dependent individuals and its ability to prevent relapse to cocaine use. Specifically, the aim of this study is to determine if memantine is superior to placebo in decreasing cocaine craving, psychological symptoms, functional impairment, and discontinuation of treatment for cocaine abuse.

Participants will enter a 2-week, single-blind, placebo lead-in phase, during which they will visit the clinic three times each week. At each study visit, urine samples and other rating assessments will be collected. In addition, participants will attend weekly therapy sessions. In order to continue in the trial, participants are required to attend at least four out of the first six study visits and both therapy sessions. Eligible participants will then be randomly assigned to receive either memantine or placebo for the duration of the 12-week, double-blind phase of the trial. Study visits will continue to occur three times each week; participants will also receive weekly therapy. Memantine will be taken twice each day. Participants who complete the 12-week trial will enter a 2-week lead-out phase, during which they will be tapered back to a placebo in a single-blind manner. Weekly psychotherapy sessions will continue until the end of Week 14.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for current cocaine dependence
* Use of cocaine at least four days in the month prior to enrollment or episodic cocaine binges of at least $200 worth at least twice each month (confirmed by urine toxicology test)

Exclusion Criteria:

* Meets DSM-IV criteria for major depression, bipolar disorder, schizophrenia, or any psychotic disorder other than transient psychosis due to drug abuse
* History of seizures in the two years prior to enrollment
* History of seizures related to current substance abuse (including cocaine, alcohol, or benzodiazepine)
* History of an allergic reaction to memantine
* Chronic organic mental disorder
* Current significant suicidal risk, history of significant suicidal behavior, or any suicide attempt within the year prior to enrollment
* Pregnant or breastfeeding
* Failure to use adequate contraception
* Unstable physical disorders that might make participation hazardous, such as hypertension, acute hepatitis (individuals with chronic mildly elevated transaminase levels at 2 to 3 times the upper normal limit are not excluded if their PT/PTT is normal), renal impairment, or diabetes
* Current coronary vascular disease, or suspected by an abnormal ECG or history of cardiac symptoms
* Cardiac conduction system disease, as indicated by QRS duration greater than 0.11
* History of failure to respond to a previous trial with memantine
* Currently meets DSM-IV criteria for substance dependence or abuse disorder other than nicotine or marijuana
* Currently taking psychotropic medications, excluding zolpidem or trazodone for insomnia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2003-03; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances R Levin, M.D., Principal Investigator — Research Foundation for Mental Hygiene, Inc.
Locations (1):
- Research Foundation for Mental Hygiene, Inc., New York, New York, United States

REFERENCES:
- See also: Substance Treatment and Abuse Research Service (STARS) — http://www.stars.columbia.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who applied for treatment at Columbia University's Substance Treatment and Research Service (STARS) outpatient clinic in New York City, USA, were recruited for this study. The study recruited from March 2003-February 2007.
Pre-assignment Details: patients entered a 2-week, single-blind placebo lead-in period. To be eligible for randomization, patients were required to attend at least 2 of 4 scheduled therapy sessions and to submit at least 4 of 6 scheduled urine samples during the two weeks of the lead-in period.
Groups:
- Memantine: Memantine 40mg/day
- Placebo: Placebo daily dose
Period: Overall Study
Arm/Group | Memantine | Placebo
Started | 39 | 42
Completed | 22 | 27
Not Completed | 17 | 15
Not completed — Lost to Follow-up | 5 | 5
Not completed — discontinued intervention | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Memantine | Placebo | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 42 | 81
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (7) | 40 (9) | 40 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 31 | 33 | 64
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81

OUTCOME MEASURES:

1. Secondary Outcome: Cocaine Abstinence Based on Daily Self Reported Cocaine Use
Description: A binary indicator of sustained abstinence, defined as three consecutive weeks of no cocaine use, obtained by self-report and verified using negative urine toxicology results, at any point of the trial;
Time Frame: reported weekly cocaine use for 12 weeks/ or study participation
Population: All analyses were performed on an intent-to-treat basis
Measure: Number; unit: participants
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 39 | 42
participants | 15 | 13

2. Primary Outcome: Weekly Cocaine Use
Description: Mean number of cocaine using days per week based on self reported use verified by cocaine toxicology results.
Time Frame: weekly use during length of study participation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Memantine | Placebo
Number analyzed (Participants) | 39 | 42
days | 1.1 (1.9) | 1.3 (1.8)

ADVERSE EVENTS:
Arm/Group | Memantine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 2/42
Other Adverse Events (participants affected / at risk) | 24/39 | 28/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=39) | Placebo (N=42)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — abdominal pain
finger fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — fingure fracture
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Memantine (N=39) | Placebo (N=42)
headache (Nervous system disorders) | 5 (5) | 7 (7) — headache
insomnia (General disorders) | 3 (3) | 6 (6) — insomnia
muscle aches (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) — muscle aches
chills (General disorders) | 0 (0) | 3 (3) — chills
fever (General disorders) | 0 (0) | 3 (3) — fever
light headed (General disorders) | 4 (4) | 3 (3) — light headed
anxiety (Psychiatric disorders) | 2 (2) | 2 (2) — anxiety
back ache (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — back ache
GI upset (Gastrointestinal disorders) | 2 (2) | 2 (2) — GI upset
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) — nausea
drowsiness (General disorders) | 3 (3) | 1 (1) — drowsiness
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — rash
diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) — diarrhea

LIMITATIONS AND CAVEATS:
participants who had achieved abstinence during the lead-in remained abstinent throughout the trial and there was little relapse-like behavior for a medication to address.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No